CLINICAL TRIAL: NCT06455852
Title: Vaccine- and Infection-derived Correlates of Protection for Cholera.
Acronym: CoP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Jason B. Harris, MD, Pediatrician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PR-24048
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cholera
MeSH Terms: conditions — Cholera | interventions — Cholera Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cholera Vaccine Arm (Experimental): The investigators will measure mucosal, memory B cell and circulating antibody responses to V. cholerae in the participants using an established immunoprofiling approach. The investigators will then identify individuals who develop V. cholerae infection over a two-year period, including those with mild and asymptomatic infection. They will use a systems-serology approach to identify CoPs in the OCV (bWC) cohort and non-OCV vaccinated control (TCV) cohort. Our approach will include cross-validation and adjustments for age, sex, and baseline immunity, to identify vaccine-induced CoPs. We will also compare the performance of these CoPs with the traditional vibriocidal titer.
  Interventions: Biological: oral cholera vaccine or typhoid conjugate vaccine
- Typhoid Vaccine Arm (Other): The investigators will compare individual CoPs and immunologic signatures in the OCV and non-cholera vaccinated (TCV) control arms which are correlated with protection. This will identify individual CoPs and immunologic signatures which distinguish protective immunity derived from natural infection with V. cholerae from immunity derived from inactivated OCV response.
  Interventions: Biological: oral cholera vaccine or typhoid conjugate vaccine

INTERVENTIONS:
Biological: oral cholera vaccine or typhoid conjugate vaccine — One group of participants will receive a 2 dose oral cholera vaccine, the other set will receive a typhoid conjugate vaccine

SUMMARY:
Background: Vibrio cholerae causes millions of cholera cases and thousands of deaths annually. Vaccines are in short supply. There is no agreement on how to introduce new vaccines or evaluate their effectiveness, and the lack of 'correlates of protection' (CoPs) against cholera is a major obstacle to vaccine development. CoPs are markers of effective immune response to vaccination. While other infectious diseases have well established CoPs, none are widely accepted for cholera.

Relevance: Lack of accepted CoPs impedes development of cholera vaccines, limiting progress toward improved vaccines, slowing the licensure of new vaccines, and contributing to the current vaccine shortage; an immediate obstacle to achieving reductions in cholera-related illness and deaths. The identification of new CoPs will speed the development of improved cholera vaccines and provide a pathway to their licensure and use.

Hypothesis: The investigators hypothesize that some individuals who receive inactivated oral cholera vaccine (OCV) will develop antibody responses which predict protection against V. cholerae infection and that specific immune responses distinguish individuals who are protected against cholera by prior natural infection from those who are protected from OCVs.

Objectives: The investigators will administer an OCV or typhoid vaccine (TCV) control and monitor antibody responses to identify better CoPs for cholera following both vaccination and natural infection.

Methods: The investigators will randomize 1219 participants; 554 participants will receive an inactivated bivalent OCV, 665 participants will receive a TCV control. The investigators will collect 12 blood samples over two-years following vaccination to measure antibodies against V. cholerae and to monitor for re-infection.

Outcome measures/variables: The endpoint of interest is V. cholerae infection after vaccination. The investigators define infection as positive culture or PCR for V. cholerae or seroconversion events observed over the 2-year follow up period.

ELIGIBILITY:
Inclusion criteria

1. Ages 2 - 80 years.
2. Informed consent from study participants and guardian in case of children (2-17 years) and assent from children aged 11-17 years.
3. Intention to participate in the study for a 2-year period.
4. No major co-morbid conditions, per the supervising clinician investigator, including underlying immunodeficiency, diabetes, liver diseases, renal disease, cardiac disease, and/or active malignancy.

Exclusion criteria

1. Suffering from diarrhoea or abdominal pain or vomiting in the past 24 hours or diarrhoea lasting for more than 2 weeks in the past 6 months.
2. History of taking another oral cholera vaccine.
3. History of taking any other live or killed enteric vaccine in the last 8 weeks.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1221 (Estimated)
Dates: Start 2025-03-02 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Vibrio cholerae infection | 2 years
  Serologic, PCR or culture evidence of infection

CONTACTS AND LOCATIONS:
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
A data sharing plan will be developed in accordance with funder regulations and institutional policies. Deidentified data will be shared upon publication of study results.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Annually updated deidentified data will be provided and datasets will be provided with any study publication